CLINICAL TRIAL: NCT06084026
Title: Measuring Physical Activity Levels and Intensity Using an ActivPal™ Accelerometer in Adult and Pediatric Populations With Neuromuscular Diseases
Brief Title: Measuring Physical Activity With ActivPal
Acronym: Activpal
Status: Recruiting | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Michio Hirano, MD, Professor of Neurology, Columbia University
Other Study IDs: AAAS6805; R01AG062401 (NIH); U54NS078059 (NIH)
Record Dates: First submitted 2023-09-26; First posted 2023-10-16 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Neuromuscular Diseases
Keywords: muscle weakness; muscle; neuromuscular
MeSH Terms: conditions — Neuromuscular Diseases; Muscle Weakness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neuromuscular Disease: Patients with confirmed neuromuscular disease
  Interventions: Other: ActivPal
- Control: Participants who do not have or are not expected to have neuromuscular disease
  Interventions: Other: ActivPal

INTERVENTIONS:
Other: ActivPal — Participants will wear the activity meter (a small button like device) on their thigh for a period of 7 days at the following time-points: baseline, 6, 12, 18, 24, 30 and 36 months. The meter will be placed on their thigh at a research visit and mailed back to the study team after 7 days.

SUMMARY:
This study measures the level of physical activity in participants with neuromuscular disorders. The patient wears a small button like meter on their leg for a period of 1 week every 6 months over a period of 3 years. Participants will also have a physical exam, six minute walk test,vital signs and questionnaires.

DETAILED DESCRIPTION:
Routine physical activity can be an important indicator of health across an individual's life span. Nonetheless, the frequency of inactivity continues to be problematic for a large number of children and adolescents. Adding to that challenge, fatigue has been described as a typical symptom of neurological diseases and disorders Consumer wearables and accelerometers are becoming increasingly popular to track physical activities and monitor health and disease progression. With the increased adoption of activity trackers comes the increased generation of valuable individual-based data. Generated data has the potential to provide detailed insights into the user's behavior and lifestyle. Although methods for objectively measuring physical activity in children and adults in naturalistic settings are well established (i.e., accelerometry), they are most widely used on healthy individuals. Due to cost and technical requirements, these technologies are limited which effects their wide-scale use. Ultimately, this undermines efforts to evaluate physical activity changes and nuances among healthy and diseased populations. This is of particular interest in rare disease populations, specifically in neuromuscular diseases, where one can study a wide range of features that can be used to monitor an individual's sleep, vertical positioning, or overall physical activity. Tracking physical activity can help provide clinicians with a more accurate disease profile and help to identify possible interventions. Collection of this data could potentially provide valuable insight into an individual's daily routines, lifestyle, and behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinically or genetically confirmed neuromuscular disorder
* Control subjects who do not have a neuromuscular disease.
* Participants at least 1 years of age.

Exclusion Criteria:

* Participant has a condition, which in the opinion of the Investigator may compromise safety
* Participant has a condition, which in the opinion of the Investigator may compromise or compliance

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with clinically or geneticallly confirmed neuromuscular disorder or controls who do not have, or are not expected to have neuromuscular disease.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Mean Activity Profile (measures time spent at various raw activity levels) | Up to 3 years
  Activity level established with Activpal meter-button like device work on thigh.

SECONDARY OUTCOMES:
Mean intensity Count (measures time spent in various actions such as rest, walking etc.) | Up to 3 years
  Fatigue level established with Activpal meter--button like device worn on thigh.

OTHER OUTCOMES:
6 minute walk test (6MWT) | Up to 3 years
  Participant walks in hallway for 6 minutes as fast as possible (no running).

CONTACTS AND LOCATIONS:
Overall Officials: Michio Hirano, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No